CLINICAL TRIAL: NCT00715507
Title: Evaluation of Drug Display in Critical Care Setting
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Noah Syroid, MS, University of Utah
Other Study IDs: 10599; 1R43GM066615-01A2 (NIH)
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Decision Making
Keywords: decision making; graphic display

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: For the phase of the study in which the utility of the graphical medication monitor is assessed, the monitor will not be shown to anesthesiologists placed in the control condition.
- 2: In the experimental condition, anesthesiologists will be shown the medication monitor to aid their expertise and decision-making.
  Interventions: Device: medication monitor

INTERVENTIONS:
Device: medication monitor — the medication monitor will aid in expertise and decision-making.
  Groups: 2

SUMMARY:
To assess the clinical utility of the graphical medication monitor, results of the anesthetics for which the display was present will be compared to the results of the anesthetics in which there was no display.

DETAILED DESCRIPTION:
This study has two objectives: First, before the medication monitor is shown to anesthesiologists in a clinical setting, the PKPD models must be validated to assess the clinical reliability of the model-based predictions for patients undergoing general anesthesia. Second, once the PKPD models have been successfully validated, presenting it to anesthesiologists during administration of anesthesia will assess the impact of the graphical medication monitor. Differences in performance and patient care will be determined by comparing anesthesiologists who are presented with the monitor to those who care for patients without the monitor.

ELIGIBILITY:
Inclusion Criteria:

* Board certified attending anesthesiologists at the University of Utah Health Sciences Center and supervised anesthesiology residents and have been trained on the graphic display

Exclusion Criteria:

* Board certified attending anesthesiologists at the University of Utah Health Sciences Center and supervised anesthesiology residents that have not been trained on the graphic display

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Board certified attending anesthesiologists at the University of Utah Health Sciences Center and supervised anesthesiology residents
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2003-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
assess differences between medication administration data and patient information with and without the use of the graphical medication monitor. | preoperative, intraoperative and postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ken Johnson, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States